CLINICAL TRIAL: NCT01564472
Title: Validation of Sleepware G3 Autoscoring Algorithm
Status: Withdrawn | Type: Observational
Why Stopped: De-identified PSGs were to be scored by a vendor prior to being sent to the sponsor. Issues occurred with vendor and no PSGs were analyzed by the sponsor.
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Other Study IDs: Dx-1152-SWGVAL-SS
Record Dates: First submitted 2012-03-20; First posted 2012-03-27 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Polysomnography Scoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PSG Scoring: Retrospective, de-identified PSG studies will be collected and scored by registered polysomnogrpahy technicians. The manually scored studies will be compared to the automatic scoring performed by the new Sleepware Software G3 Autoscoring Algorithm.
  Interventions: Other: PSG Scoring

INTERVENTIONS:
Other: PSG Scoring — No participants will be enrolled and no interventions, besides PSG scoring will be utilized.

SUMMARY:
The objective of this study is to validate the ability of the Sleepware G3 polysomnography software platform to correctly identify and score sleep related events.

ELIGIBILITY:
Inclusion Criteria:

* AASM Compliant PSG studies

Exclusion Criteria:

* NA

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any retrospective, de-identified adult polysomnogram collected using American Society of Sleep Medicine (AASM) criteria.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
PSG Scoring Validity | 6 months
  The objective of this study is to validate the ability of the Sleepware G3 polysomnography software platform to correctly identify and score sleep related events. Specifically, the study will compare Sleepware autoscoring of respiratory events, sleep staging, leg movements, micro-arousals and desaturations, among possible others events, to manual scoring by two registered polysomnographic technologists (RPSGT).